CLINICAL TRIAL: NCT02922868
Title: Assessment of Infection Control, Practice Efficiency, and Health Economics of Sheathed Versus Standard Flexible Cystoscopy
Brief Title: Assessment of Infection Control, Practice Efficiency, and Health Economics of Sheathed Versus Standard Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Cogenix Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00036203
Record Dates: First submitted 2016-09-02; First posted 2016-10-04 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Bacteriuria
Keywords: Cystoscopy; EndoSheath; Infection Control; Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EndoSheath CST-5000 Scope (Experimental): Cogentix Medical CST-5000 Flexible Video Cystoscope with Slide-On® EndoSheath® Technology. EndoSheath CST-5000 Scope.
  Interventions: Device: EndoSheath CST-5000 Scope
- Olympus Visera Elite OTV-S190 Scope (Active Comparator): Olympus HD Flexible Cysto-Nephro Videoscope (CYF-VH) with Olympus Visera Elite Platform, including OTV-S190 Video Processor CLV-S190 Xenon Light Source. Olympus Visera Elite OTV-S190 Scope.
  Interventions: Device: Olympus Visera Elite OTV-S190 Scope

INTERVENTIONS:
Device: EndoSheath CST-5000 Scope — Cystoscopic procedures will be performed using the EndoSheath CST-5000 Scope.
  Arms: EndoSheath CST-5000 Scope
Device: Olympus Visera Elite OTV-S190 Scope — Cystoscopic procedures will be performed using the Olympus Visera Elite OTV-S190 Scope
  Arms: Olympus Visera Elite OTV-S190 Scope

SUMMARY:
The purpose of this research study is to compare the effectiveness and efficiency of using a sterile sheath (EndoSheath®) during cystoscopy versus a standard scope.

DETAILED DESCRIPTION:
The increasing costs in health care and enhanced infection control requirements necessitate the efficient and reliable use of frequently used techniques like cystoscopy. The health economics of cystoscopy are dependent on maintaining low levels of post-cystoscopy sequelae like urinary tract infection (UTI) and its potential precursors, significant asymptomatic bacteriuria and leukocytosis. Another key component of the economics and efficiency of cystoscopy is the time and cost related to the reprocessing of these devices in preparation for re-use. The use of disposable endoscope sheaths may limit the need for high level disinfection (HLD) between procedures and reduce reprocessing time and potentially prolong the cystoscope lifespan. The rationale for this study is to determine if a sheathed cystoscopy system would provide the desired cost and efficiency advantages compared to procedures done with non-sheathed cystoscopes. This is a prospective, randomized, parallel group, single center clinical trial to assess the clinical outcomes, practice efficiency and health economics of the use of sheathed cystoscopes (EndoSheath® System) compared to using standard (non-sheathed) cystoscopes. The study will evaluate the infection control (via the change in bacteriuria), clinical practice efficiency and costs of the EndoSheath technology with CST 5000 scope compared to standard cystoscopy with Olympus Visera Elite OTV-S190 digital flexible scope. There will be 30 subjects in the control group undergoing cystoscopy with the standard scope at the clinic, the Olympus Visera Elite, and 30 subjects in the study group undergoing cystoscopy with the EndoSheath system. The study is designed as a prospective, randomized controlled trial. There will be no active blinding of clinicians or subjects; however, it is anticipated that most subjects will be unaware of differences in the cystoscopy equipment that will be utilized in their routine procedures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years of age or older
* Patients undergoing de novo or follow up diagnostic or therapeutic cystoscopy procedures in a Urology clinic setting
* Antibiotic-free for at least 7 days prior to cystoscopy procedure
* Patients willing to return to the clinic at approximately two weeks (10 -14 days) post-procedure for a urine test

Exclusion Criteria:

* Patients with significant lower urinary tract obstruction, gross hematuria
* Patients having an acute pelvic inflammatory disease or symptomatic UTI
* Patients with urethral strictures
* Patients with chronic pain conditions
* Patients unwilling to return to the clinic at approximately two weeks (10 -14 days) for a urine test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gopal H Badlani, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health - Department of Urology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Post-Procedure Bacteriuria
Description: The primary endpoint will be the change in bacteriuria pre- and post-procedure between EndoSheath CST-5000 cystoscope and standard (non-sheathed) Olympus Visera Elite OTV-S190 cystoscope during the course of routine clinical use in a urology clinic. The pre-procedure measurement of bacteriuria will occur on the day of the procedure. The post-procedure measurement of bacteriuria will occur approximately two weeks (10-14 days) post-procedure. This will be assessed by urine culture exams.
Time Frame: 10-14 Days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
Participants | 0 | 1

2. Secondary Outcome: Number of Cystoscopes With Positive Bioburden Post-procedure.
Description: Immediately after completion of each cystoscopy procedure, the bioburden on the cystoscopes will be evaluated. The flexible cystoscope sheath was removed for bioburden assessment. For each cystoscope, whether sheathed or standard, two locations were assessed - the control body and the shaft. Cultures were obtained wiping the entire surface with sterile saline pledgets. The sample pledgets were placed in 1 ml sterile saline and shaken for 30 seconds. Ten drops of 0.02 ml aliquots from the sample were spotted on two 5% blood agar plates and incubated at 35°C in CO2.
Time Frame: Immediately after cystoscopy.
Measure: Number; unit: bioburdens
Units Other Than Participants: cystoscope locations
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
Number analyzed (cystoscope locations) | 30 | 30
bioburdens
  Shaft | 0 | 4
  Body | 0 | 0

3. Secondary Outcome: Total Time to Reprocess a Cystoscope
Description: The total time required for a cystoscope to be reprocessed so that it is available for re-use in a subsequent procedure will be measured.
Time Frame: Beginning from the time a cystoscope is withdrawn from the urethral meatus at the end of a procedure until the completion of reprocessing, approximately 3,869 seconds
Measure: Mean (Standard Error); unit: seconds
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
seconds | 270.91 (190) | 3838.78 (1270)

4. Secondary Outcome: Subject Assessment of Procedure.
Description: After undergoing cystoscopy, patients will be asked to complete Visual Analog Scales (VAS) instruments to determine their level of pain experienced during cystoscopy as well as their perception of discomfort with the procedure. The score range is 0 to 100. Higher scores denotes worse outcomes.
Time Frame: Approximately 2 min after the end of procedure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
units on a scale
  VAS Pain | 29.3 (23) | 26.5 (20.77)
  VAS Discomfort | 30.79 (21.41) | 29.2 (17.57)

5. Secondary Outcome: Staff Assessment of Cystoscope Reprocessing.
Description: At the end of each day while the study is in progress, 6 members of the medical staff directly involved with the reprocessing of cystoscopes will evaluate the ease of reprocessing based on a 5-point Likert scale for the following parameters: ease of Insertion, ease of manipulation, optical quality, overall ease of use. The score range is 0 to 5. Higher score denotes better outcomes. A single value was derived per staff member and summarized for the group as a whole during 6 months.
Time Frame: At the end of day of each procedure during 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
units on a scale
  Ease of Insertion | 4.27 (0.76) | 4.72 (0.55)
  Ease of Manipulation | 4.13 (0.83) | 4.5 (0.8)
  Optical Quality | 3.9 (1.15) | 4.3 (1.12)
  Overall Ease of Use | 4.02 (0.93) | 4.45 (0.85)

6. Secondary Outcome: Total Cost of Cystoscopy Reprocessing
Description: The health economics of reprocessing will be evaluated by associating personnel hourly costs with cystoscope reprocessing time segments. The total cost was averaged between pre-cleaning, cleaning, disinfection, rinsing, and drying for the 30 cystoscopes in each group for a duration of 6 months.
Time Frame: 6 months
Measure: Number; unit: Dollars
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
Dollars | 57,000.00 | 32,000.00

7. Secondary Outcome: Number of Procedures Per Day Per Scope.
Description: Number of procedures per day per scope. On a daily basis urology outpatient clinic performs an average of 5 cystoscopies.
Time Frame: Per day.
Measure: Mean (Standard Deviation); unit: Number of procedures per day per scope
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Number analyzed (Participants) | 30 | 30
Number of procedures per day per scope | 5 (2) | 5 (2)

ADVERSE EVENTS:
Time Frame: 15 days after procedure
Arm/Group | EndoSheath CST-5000 Scope | Olympus Visera Elite OTV-S190 Scope
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes